CLINICAL TRIAL: NCT06162572
Title: A Phase 1b/2, Multicenter, Open-label Platform Study of Select Immunotherapy Combinations in Adult Participants With Previously Untreated Advanced Non-small Cell Lung Cancer (NSCLC) With High PD-L1 Expression
Brief Title: Phase 1b/2 Platform Study of Select Immunotherapy Combinations in Participants With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPLFIO-174
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- S095018 (anti-TIM3 antibody) in combination with cemiplimab (Experimental): Part A: Combination-therapy safety lead-in
  Interventions: Drug: S095018; Drug: Cemiplimab
- S095024 (anti-CD73 antibody) in combination with cemiplimab (Experimental): Part A: Combination-therapy safety lead-in
  Interventions: Drug: S095024; Drug: Cemiplimab
- S095029 (anti-NKG2A antibody) in combination with cemiplimab (Experimental): Part A: Combination-therapy safety lead-in
  Interventions: Drug: S095029; Drug: Cemiplimab
- S095018 (anti-TIM3 antibody) RDE in combination with cemiplimab (Experimental): Part B: Randomized dose expansion
  Interventions: Drug: S095018 Recommended Dose Expansion (RDE); Drug: Cemiplimab
- S095024 (anti-CD73 antibody) RDE in combination with cemiplimab (Experimental): Part B: Randomized dose expansion
  Interventions: Drug: S095024 RDE; Drug: Cemiplimab
- S095029 (anti-NKG2A antibody) RDE in combination with cemiplimab (Experimental): Part B: Randomized dose expansion
  Interventions: Drug: S095029 RDE; Drug: Cemiplimab
- Cemiplimab (control arm) (Active Comparator): Part B: Randomized dose expansion
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: S095018 — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095018 (anti-TIM3 antibody) in combination with cemiplimab
Drug: S095024 — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095024 (anti-CD73 antibody) in combination with cemiplimab
Drug: S095029 — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095029 (anti-NKG2A antibody) in combination with cemiplimab
Drug: S095018 Recommended Dose Expansion (RDE) — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095018 (anti-TIM3 antibody) RDE in combination with cemiplimab
Drug: S095024 RDE — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095024 (anti-CD73 antibody) RDE in combination with cemiplimab
Drug: S095029 RDE — Via IV infusion on Day 1 of each 21-day cycle
  Arms: S095029 (anti-NKG2A antibody) RDE in combination with cemiplimab
Drug: Cemiplimab — 350 mg via IV infusion on Day 1 of each 21-day cycle

SUMMARY:
This is a Phase 1b/2 study evaluating the anti-PD1 antibody, cemiplimab, in combination with either S095018 (anti-TIM3 antibody), S095024 (anti-CD73 antibody), or S095029 (anti-NKG2A antibody) in adult participants with previously untreated advanced/metastatic non-small cell lung cancer (NSCLC) with high PD-L1 expression. The study includes two parts: part A, the combination-therapy safety lead-in phase to determine the recommended dose for expansion (RDE) for S095018, S095024, and S095029 in combination with cemiplimab and part B, the randomized dose expansion phase to assess the efficacy of S095018, S095024, or S095029 in combination with cemiplimab. Study treatment will be administered for a maximum of 108 weeks, or until confirmed disease progression per iRECIST and/ or until meeting other treatment discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥ 18 years
* Written informed consent
* Histologically (squamous or non-squamous) or cytologically documented locally advanced NSCLC not eligible for surgical resection and/or definitive chemoradiation, or metastatic NSCLC
* No prior systemic treatment for locally advanced or metastatic NSCLC
* High tumor cell PD-L1 expression [Tumor Proportion Score (TPS) ≥50%] based on documented status as determined by an approved test
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Measurable disease as determined by RECIST v1.1

Exclusion Criteria:

* Tumors harboring driver mutations/genetic aberrations for which targeted therapies are approved as frontline treatment (e.g. EGFR mutation, ALK fusion oncogene, ROS1 aberrations)
* Prior immune checkpoint inhibitor therapy
* Active brain metastases
* Participants with active and uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Uncontrolled HIV infection. Participants with HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are allowed to enroll
* Active, known or suspected autoimmune disease or immune deficiency
* History of hypersensitivity reactions to any ingredient of the investigational medicinal product (IMP) and other monoclonal antibody (mAbs) and/or their excipients
* History of interstitial lung disease, idiopathic pulmonary fibrosis, drug-induced pneumonitis, idiopathic pneumonitis or active pneumonitis ≥ grade 2
* History of inflammatory bowel disease or colitis ≥ grade 2
* History of hemophagocytic lymphohistiocytosis.
* Systemic chronic steroid therapy (>10mg/d prednisone or equivalent)
* Clinically significant infection, as assessed by the investigator
* Pregnant or breast-feeding (lactating) women
* Participants with a history of allogeneic organ transplantation (e.g., stem cell or solid organ transplant)
* Any medical condition that would in the investigator's judgement prevent the participant's participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) during the first 2 cycles of combination treatment | Through the end of the Cycle 2 (each cycle is 21 days)
  Part A
Incidence and severity of adverse events (AEs) | From the signed informed consent form (ICF) to 30 days after the last dose
  Part A
Incidence and severity of serious adverse events (SAEs) | From the signed ICF to 120 days after the last dose
  Part A
Adverse Events (AEs) Leading to Dose Interruption, Modification, or Delays | From signed ICF through treatment discontinuation (up to 108 weeks of treatment)
  Part A
Adverse Events (AEs) Leading to Permanent Treatment Discontinuation | From signed ICF through treatment discontinuation (up to 108 weeks of treatment)
  Part A
Objective Response (OR) | Until study termination (approximately 2 years)
  Part B: Participants who achieve complete response (CR) or partial response (PR), as per investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Objective Response (OR) | Until study termination (approximately 3 years)
  Part A: Participants who achieve CR or PR, as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST) as assessed by the investigator.
Best Overall Response (BOR) | Until study termination (approximately 3 years)
  Part A and B: The best response designation using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST), recorded between the date of the first dose of treatment and the date of the first objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. CR or PR used in the BOR requires a confirmation that is at least 4 weeks apart.
Duration of Response (DoR) | Until study termination (approximately 3 years)
  Part A and B: The time from the first documentation of CR or PR until the documented progressive disease (PD) or death, as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST) as assessed by the investigator.
Disease Control (DC) | Until study termination (approximately 3 years)
  Part A and B: Participants who achieved stable disease (SD), PR, or CR (based on participant's best response), as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST) as assessed by the investigator.
6-month Durable Response (6-month DR) | Until study termination (approximately 3 years)
  Part A and B: Continuous CR or PR for ≥ 6 months, recorded between the date of the first dose of treatment and the date of the first objectively documented progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or the date of subsequent anti-cancer therapy, whichever occurs first.
Progression-Free Survival (PFS) | Until study termination (approximately 3 years)
  Part A and B: The time from the first dose to the first documented PD or death due to any cause, whichever occurs first, as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST) as assessed by the investigator.
Plasma or serum concentration of S095018 | From first dose to 30 days after the last dose
  Part A and B
Plasma or serum concentration of S095024 | From first dose to 30 days after the last dose
  Part A and B
Plasma or serum concentration of S095029 | From first dose to 30 days after the last dose
  Part A and B
Incidence and titer of anti-drug antibodies (ADA) directed against S095018 | From screening to 90 days after the last dose
  Part A and B
Incidence and titer of anti-drug antibodies (ADA) directed against S095024 | From screening to 90 days after the last dose
  Part A and B
Incidence and titer of anti-drug antibodies (ADA) directed against S095029 | From screening to 90 days after the last dose
  Part A and B
Incidence and severity of adverse events (AEs) | From signed ICF to 30 days after the last dose
  Part B
Incidence and severity of serious adverse events (SAEs) | From signed ICF to 120 days after the last dose
  Part B
Adverse Events (AEs) Leading to Dose Interruption, Modification, or Delays | From signed ICF through treatment discontinuation (up to 108 weeks of treatment)
  Part B
Adverse Events (AEs) Leading to Permanent Treatment Discontinuation | From signed ICF through treatment discontinuation (up to 108 weeks of treatment)
  Part B

CONTACTS AND LOCATIONS:
Locations (73):
- United States (7):
  - Loma Linda University, Loma Linda, California
  - University of Kansas Medical Center, Lawrence, Kansas
  - Henry Ford Health, Detroit, Michigan
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia
- Argentina (2):
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Sanatorio Parque S.A., Santa Fe
- Australia (4):
  - Border Medical Oncology Research Unit, Albury
  - Flinders Medical Centre, Bedford Park
  - Sunshine Hospital, St Albans
  - Latrobe Regional Health, Traralgon
- Austria (3):
  - Ordensklinikum Linz Elisabethinen, Linz
  - Universitatsklinikum St. Poelten, Sankt Pölten
  - Medical University of Vienna - Akh, Vienna
- Belgium (2):
  - Jessa Ziekenhuis, Hasselt
  - Uz Leuven Campus Gasthuisberg, Leuven
- Brazil (13):
  - Hospital de Amor - Barretos, Barretos
  - Supera Oncologia, Chapecó
  - CIONC, Curitiba
  - ONCOSITE, Ijuí
  - Liga Contra O Cancer - Natal, Natal
  - Santa Casa de Porto Alegre, Porto Alegre
  - Hospital São Lucas Da Pucrs, Porto Alegre
  - Oncoclinicas Rj, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital A C Camargo, São Paulo
  - Hospital São Camilo, São Paulo
  - Oncoclinicas Sp, São Paulo
  - Hospital Albert Einstein, São Paulo
- France (5):
  - Centre Georges Francois Leclerc, Dijon
  - Chu Grenoble Alpes, Grenoble
  - Institut Paoli Calmette, Marseille
  - Centre René Gauducheau/Inst de Cancér. de L'Ouest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Hong Kong (3):
  - Hong Kong United Onology Centre, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (3):
  - Farkasgyepu Tudogyogyintezet, Farkasgyepű
  - Bugat Pal Hospital, Gyöngyös
  - Pecsi Tudomanyegyetem, Klinikai Kozpont, Pécs
- Italy (9):
  - Centro Di Riferimento Oncologico, Aviano
  - Inst. Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Irccs Fondazione Istituto Nazionale Dei Tumori, Milan
  - Istituto Europeo Di Oncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ist. Nazionale Tumori Irccs Fondazione G Pascale, Napoli
  - Azienda Ospedaliera S. Maria Della Misericordia, Perugia
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas I.R.C.C.S, Rozzano
- Romania (4):
  - Inst Oncologic "Prof Dr I Chiricuta" Cluj Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie, Craiova
  - Centrul de Radioterapie Amethyst, Otopeni
  - Ploiesti Municipal Hospital, Ploieşti
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Gacheon University Gil Medical Center, Incheon
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Vall D' Hebron Institute of Oncology (Vhio), University Hospital, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clinica Universitaria de Navarra (Madrid), Madrid
  - Hospital Univ. Hm Sanchinarro Start Ciocc Early Phase, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Clinica Universitaria de Navarra (Pamplona), Pamplona
  - Hospital Virgen Del Rocío, Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (4):
  - The Royal Marsden in Sutton, London
  - The Royal Marsden in Chelsea, London
  - Imperial College London, London
  - The Christie Nhs Foundation Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/